CLINICAL TRIAL: NCT00002169
Title: A Phase II, Randomized, Placebo-Controlled Study to Determine the Effects of Viracept on the Clinical Outcome of Cytomegalovirus (CMV) Retinitis in AIDS Patients Who Are Receiving Standard Induction and Maintenance Therapy for This Infection
Brief Title: A Study of Viracept in AIDS Patients With Cytomegalovirus Retinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 259A; Study 517; AG1343-517
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Placebos; Antiviral Agents; Cytomegalovirus Retinitis; Treatment Outcome; Nelfinavir
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if it is safe and effective to give Viracept to AIDS patients who are already being treated for cytomegalovirus (CMV) retinitis.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Newly diagnosed or first progression of CMV retinitis.

Exclusion Criteria

Prior Medication:

Excluded:

Prior therapy (or less than 2 weeks) with protease inhibitor other than saquinavir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Univ of Southern California / LA County USC Med Cntr, Los Angeles, California
  - Univ of California / UCI Med Ctr, Orange, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Harbor UCLA Med Ctr, Torrance, California
  - George Washington Univ, Washington D.C., District of Columbia
  - Northwestern Univ / SOCA, Chicago, Illinois
  - Univ of Texas Med Branch, Galveston, Texas
  - Baylor Univ, Houston, Texas